CLINICAL TRIAL: NCT01471301
Title: Ultrasound Evaluation of Hands in Patients With Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Leticia Pirozzi Buosi, Ultrasound evaluation of hands in patients with Systemic Lupus Erythematosus, Federal University of São Paulo
Other Study IDs: ABuosi
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Lupus Erythematosus, Systemic; Arthritis, Rheumatoid
Keywords: systemic lupus erythematosus; rheumatoid arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate ultrasound hands in patients with systemic lupus erythematosus.

DETAILED DESCRIPTION:
Introduction: The systemic lupus erythematosus (SLE) is a disease with a common articular involvement. Approximately 1-2% of patients with SLE have joint inflammation similar to rheumatoid arthritis (RA). There are no well-designed studies of lupus arthropathy.

Primary objectives: To evaluate the ultrasonographic examination of the hands in patients with systemic lupus erythematosus and make its correlation with examination of patients with rheumatoid arthritis (RA) established and with clinical, serological, radiological and functional.

Material and methods: a transversal study will be carried out on patients diagnosed with with SLE and RA.

Clinical Instruments: count of swollen and tender joints, visual analogue scale (VAS) for pain (0-10 cm), edema and for disease activity; disease activity (DAS 28 and SLEDAI), hand grip strength and pinch (Jamar dynamometer and Preston Pinch Gauge); functional questionnaires (HAQ and DASH). It will be observed the presence of "puffy hands", Raynaud's phenomenon and presence of autoantibodies.

Radiographic instruments: evaluation of radiographs of hands and wrists according to the Sharp score modified by van der Heijde. Ultrasonographic Instruments (quantitative and semi-quantitative measures): synovial hyperplasia, synovial blood flow (Power Doppler), bone erosions and cartilage. The joints that will be evaluated: radiocarpal, distal radioulnar, first to fifth metacarpophalangeal and proximal interphalangeal. Ultrasonographic interobserver reproducibility will be carried out in 10% of the patients. All the examinators will be blind for each other findings. Rheumatoid factor and anti-CCP will be investigated in RA patients. Statistical significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years;
* female and male;
* patients with SLE, according to the revised classification criteria of the ACR (Arthritis Rheum, 1997) with current or previous joint activity (arthritis or arthralgia;
* patients with established RA according to ACR classification criteria (Arthritis Rheum, 1988)

Exclusion Criteria:

* changing the dose or drug-based immunosuppression in the last 3 months.
* corticosteroid pulse therapy in the last 30 days;
* infiltration with corticosteroids at hand in the last 3 months;
* previous surgery in the joints studied;
* irreducible deformity of the joints studied;
* overlap with other joint diseases or collagen;
* chiropractic diabetic;
* hypothyroidism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ambulatory rheumatology
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Letícia Pirozzi Buosi, Principal Investigator — Outros
Locations (1):
- Unifesp, São Paulo, São Paulo, Brazil